CLINICAL TRIAL: NCT04132245
Title: Famil-based Obesity Prevention Trial in Latino Families
Brief Title: Family-based Outcome Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Dr. Fitzgibbon, Professor, Dept. of Medicine and School of Public Health, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21CA121423 (NIH)
Record Dates: First submitted 2016-05-16; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Obesity
Keywords: childhood obesity; minorities; diet; physical activity; parents
MeSH Terms: conditions — Obesity; Pediatric Obesity; Motor Activity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- obesity prevention (Experimental): Families were randomized to an obesity prevention intervention arm or a general health control arm.
  Interventions: Behavioral: Obesity prevention intervention trial
- behavioral intervention (Experimental): there are two arms in this study. An active intervention arm and a control arm
  Interventions: Behavioral: behavioral intervention

INTERVENTIONS:
Behavioral: behavioral intervention — Families were randomized to a 14-week family based obesity prevention intervention or a 14-week general health intervention
  Arms: behavioral intervention
Behavioral: Obesity prevention intervention trial — Families were randomized to a 14-week obesity prevention intervention or a 14-week general health intervention
  Arms: obesity prevention

SUMMARY:
Many obesity related risk factors are strikingly apparent in minority populations. Mexican-American children have the highest rates of overweight. The goals of this study are to: 1) test the acceptability of a 14-week family-based intervention with 3-5 year old children and their parents; 2) Estimate the effectiveness of a 14-week family-based intervention designed to show smaller changes, on average, in BMI appropriate for growth; 3) estimate the effectiveness of a 14-week family-based intervention designed to produce changes in television viewing, physical activity, fat, fiber, and fruit and vegetable intake in 3-5 year old Latino children and their parents at post-intervention and Year 1 follow-up.

ELIGIBILITY:
Inclusion Criteria:

* have received an annual physical
* parent or guardian willing to give consent
* parent or guardian willing to provide demographic and anthropometric data and agree to complete food intake and physical activity information for their child

Exclusion Criteria:

* requires a specialized diet outside of that served by the Chicago Public Schools
* has a chronic physical or behavioral disorder that requyires participant to be under close emdical psychologicagl supervision and routinely absent from the study

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Body mass index | 1 year
  we measured the change in BMI of the children at baseline and post-intervention